CLINICAL TRIAL: NCT01558531
Title: Drug Eluting Balloon in peripherAl inTErvention for In-Stent Restenosis: the DEBATE-ISR Study
Brief Title: Drug Eluting Balloon in Peripheral Intervention for In-Stent Restenosis
Acronym: DEBATE-ISR
Status: Suspended | Type: Observational
Why Stopped: slow enrollment
Sponsor: Leonardo Bolognese, MD (Other)
Responsible Party: Sponsor-Investigator, Leonardo Bolognese, MD, Director, Ospedale San Donato
Organization: Ospedale San Donato (Other)
Other Study IDs: Arezzo006
Record Dates: First submitted 2012-03-17; First posted 2012-03-20 (Estimated); Last update posted 2015-02-03 (Estimated); Status verified 2015-02

CONDITIONS: Peripheral Arterial Disease
Keywords: peripheral arterial disease; drug-eluting balloon; restenosis
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- DEB: paclitaxel-eluting balloon angioplasty
  Interventions: Device: DEB
- conventional PTA: historical conventional balloon angioplasty control group (patients referred to our institution between 2008 and 2009)
  Interventions: Device: POBA

INTERVENTIONS:
Device: DEB — paclitaxel-eluting balloon angioplasty
  Groups: DEB
Device: POBA — conventional balloon angioplasty
  Groups: conventional PTA

SUMMARY:
The purpose of this study is to evaluate the efficacy of drug-eluting balloon angioplasty followed versus conventional balloon angioplasty in superficial femoral artery and popliteal artery re-stenosis.

ELIGIBILITY:
Inclusion Criteria:

* age>18 years
* intermittent claudication (Fontane III or IV)
* angiographic stenosis>50% or occlusion of superficial femoral-popliteal artery>40mm, previously treated with nitinol stent implantation, with at least one below-knee vessel to the ankle

Exclusion Criteria:

* allergy to Paclitaxel
* contraindication for combined antiplatelet treatment
* life expectancy <1 year
* hypersensitivity or contraindication to one of the study drugs
* lack of consent
* need for amputation
* angiographic evidence of stent fracture

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients referring to our institution for peripheral artery disease
Sampling Method: Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2010-01; Primary Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
angiographic binary re-restenosis | 12 months
  incidence of angiographic binary re-restenosis

SECONDARY OUTCOMES:
major amputation | 24 months
  incidence of major amputation
stent thrombosis | 24 months
  incidence of stent thrombosis
target lesion revascularization | 24 months
  incidence of target lesion revascularization

CONTACTS AND LOCATIONS:
Locations (1):
- Cardiovascular Department, Ospedale S.Donato, Arezzo, AR, Italy

REFERENCES:
- [Derived] Grotti S, Liistro F, Angioli P, Ducci K, Falsini G, Porto I, Ricci L, Ventoruzzo G, Turini F, Bellandi G, Bolognese L. Paclitaxel-Eluting Balloon vs Standard Angioplasty to Reduce Restenosis in Diabetic Patients With In-Stent Restenosis of the Superficial Femoral and Proximal Popliteal Arteries: Three-Year Results of the DEBATE-ISR Study. J Endovasc Ther. 2016 Feb;23(1):52-7. doi: 10.1177/1526602815614555. Epub 2015 Oct 28. PMID 26511896
- [Derived] Liistro F, Angioli P, Porto I, Ricci L, Ducci K, Grotti S, Falsini G, Ventoruzzo G, Turini F, Bellandi G, Bolognese L. Paclitaxel-eluting balloon vs. standard angioplasty to reduce recurrent restenosis in diabetic patients with in-stent restenosis of the superficial femoral and proximal popliteal arteries: the DEBATE-ISR study. J Endovasc Ther. 2014 Feb;21(1):1-8. doi: 10.1583/13-4420R.1. PMID 24502477